CLINICAL TRIAL: NCT06535295
Title: Comparison of Physical Activity, Functional Capacity and Quality of Life Between Older Patients With Chronic Comorbidities and Healthy Peers
Brief Title: Physical Activity, Functional Capacity and Quality of Life in Older Patients With Chronic Comorbidities
Status: Completed | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, Hikmet Ucgun, Assistant Professor, Biruni University
Other Study IDs: auhucgun02
Record Dates: First submitted 2024-07-25; First posted 2024-08-02 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Obesity; Hypertension; Type 2 Diabetes
Keywords: Physical Activity; Functional Capacity; Quality of Life
MeSH Terms: conditions — Obesity; Hypertension; Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Obesity Group: Older patients with obesity
- Hypertension Group: Older patients with hypertension
- Type 2 Diabetes Group: Older patients with type 2 diabetes
- Healthy Group: Healthy older adults

SUMMARY:
The prevalence of obesity, hypertension (HT) and type 2 diabetes (T2D) is increasing. The adoption of an increasingly sedentary lifestyle is one of the main factors contributing to the increased incidence of chronic diseases such as obesity, cardiovascular diseases, HT and T2D. Furthermore, lack of physical activity leads to a decline in functional capacity in these individuals, which facilitates the progression of HTN, T2D and obesity. The presence of multiple chronic comorbidities can exacerbate the negative impact on health-related quality of life. The main aim of this study was to compare the levels of physical activity, functional capacity and quality of life between elderly individuals with chronic comorbidities such as HTN, T2D and obesity and their healthy peers. Quality of life, functional capacity , and physical activity level will be assessed by SF-36 questionnaire, 6-minute walk test, and the International Physical Activity Questionnaire-short form, respectively.

DETAILED DESCRIPTION:
Globally, the elderly population is increasing, along with a significant rise in the prevalence of chronic conditions such as obesity, hypertension (HT) and type 2 diabetes (T2D). The World Health Organization (WHO) reported in 2021 that over 2 billion adults were overweight, with more than 800 million classified as obese. At the same time, HT affected 1.28 billion adults globally, and the incidence of T2D surged from 108 million in 1980 to 537 million in 2021. Focusing on the older population, recent studies show that around 50% of older adults are affected by obesity, approximately 52.9% suffer from HT, and about 27.5% have T2D. The high prevalence of chronic diseases among older adults poses a significant health challenge and strains healthcare systems globally. This challenge is driven by increased life expectancy and the rapid aging of the population, which together lead to a larger elderly population and, consequently, a higher incidence of chronic diseases.

Obesity, T2D, and HT can lead to complications in the cardiovascular and musculoskeletal systems, which in turn are likely to negatively affect PA, functional capacity, and QoL. For instance, obesity can increase the load on joints due to excessive weight, thereby restricting mobility, while T2D may adversely affect walking capacity through peripheral neuropathy and vascular complications. Hypertension could exacerbate symptoms during PA by increasing the cardiovascular load. In managing chronic diseases such as obesity, HT, and T2D, medications play a vital role in controlling these conditions and preventing complications. Nevertheless, even with this treatment, patients may continue to experience declines in functional capacity, PA, and QoL. The impact of chronic diseases such as obesity, HT, and T2D on PA, functional capacity, and QoL in older adults remains unclear in the literature. Although early detection and prevention of these conditions are important, the specific effects on these health aspects are not well-defined. Research indicates that while these conditions can influence health, their impact varies among individuals, and effective management may mitigate some adverse effects. Further research is needed to clarify how chronic diseases such as obesity, HT, and T2D affect PA, functional capacity, and QoL in the older population, as there remains a significant gap in empirical data regarding these effects.

Therefore, the aim of our study is to compare PA, functional capacity, and QoL between patients with obesity, HT, T2D, and healthy controls, and to elucidate the differing impacts of these chronic conditions on these parameters. The physical activity level will be evaluated using the short form of the International Physical Activity Questionnaire (IPAQ), the functional capacity will be evaluated using the 6-minute walk test, and the quality of life will be evaluated using the SF-36 Quality of Life Scale. At the end of the study, physical activity, functional capacity and quality of life will be compared between older patients with chronic comorbidities and healthy peers.

ELIGIBILITY:
Inclusion Criteria of Patients with Obesity:

* Being 65 years of age or older
* Body Mass Index (BMI) ≥30 kg/m²

Inclusion Criteria of Patients with Hypertension:

* Being 65 years of age or older
* Being diagnosed with hypertension
* Regular use of antihypertensive medication

Inclusion Criteria of Patients with Type 2 Diabetes:

* Being 65 years of age or older
* Being diagnosed with type 2 diabetes
* HbA1c levels: 57-78 mmol/mol (IFCC) or 7.4-9.3% (NGSP)

Inclusion Criteria of Healthy Older Adults:

* Being 65 years of age or older
* Not having any chronic condition diagnosis

Exclusion Criteria:

* History of unstable angina or myocardial infarction
* Having a poor glycemic control
* Having a diabetic neuropathy
* Having a lower extremity musculoskeletal problem
* Having a balance disorder condition
* Having a cognitive impairment

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Thirty-seven patients with obesity Thirty-seven patients with hypertension Thirty-seven patients with type 2 diabetes Thirty-seven healthy older adults
Sampling Method: Probability Sample
Enrollment: 148 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Level of Physical Activity | 10-15 minutes
  Physical activity will be assessed by SF-36 questionnaire. The SF-36 consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Level of Functional Capacity | 15-20 minutes
  The 6-minute walking test will be used to assess the functional capacity. Participants will be recorded in a 30-meter straight corridor for 6 minutes at their own walking speed, as fast as possible but without running. The walking distance will be recorded in meters.
Level of Quality of Life | 8-10 minutes
  Quality of life will be assessed by the International Physical Activity Questionnaire-short form. (IPAQ-SF). The IPAQ scoring protocol assigns the following MET values to walking, moderate, and vigorous intensity activity: 3.3 METs, 4.0 METs, and 8.0 METs, respectively. If the participants reported at least 150 min/wk of walking, moderate, or vigorous intensity physical activity.

CONTACTS AND LOCATIONS:
Overall Officials: Hikmet Ucgun, PT, PhD, Principal Investigator — Atlas University
Locations (1):
- Istanbul Atlas University, Istanbul, Kaguthane, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No